CLINICAL TRIAL: NCT04552951
Title: Estudio Destinado a Valorar la Utilidad de Vitamina D Sobre Morbilidad y Mortalidad de la infección Por Virus SARS-COV-2 (COVID-19) en el Hospital Universitario Central de Asturias
Brief Title: Effect of Vitamin D on Morbidity and Mortality of the COVID-19
Acronym: COVID-VIT-D
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación para la Investigación Biosanitaria del Principado de Asturias (Other)
Collaborators: Hospital Universitario Central de Asturias (Other); Instituto de Investigación Sanitaria del Principado de Asturias (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-019-PF-CAANJ
Record Dates: First submitted 2020-05-21; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Intervention Model Description: Patients receiving any form. of vitamin D excluded from the study. Randomized study (Initial serum calcidiol levels blinded )
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Receiving 1 dose of 100.000 iu of Cholecalciferol when the COVID 19 Disease is diagnosed
  Interventions: Drug: Cholecalciferol
- Control (No Intervention): No vitamin D

INTERVENTIONS:
Drug: Cholecalciferol — Single doe of 100.000 IU
  Other Names: Vitamin D
  Arms: Active

SUMMARY:
Patients diagnosed of COVID-19 disease are randomized to receive a single dose of 100.000 IU of Cholecalciferol (Vitamin D arm) or no vitamin D (on top of the current medication used to treat COVID 19).

Clinical, radiological and biochemical outcomes of COVID 19 disease as well as mortality are evaluated.

DETAILED DESCRIPTION:
Efficacy parameters to compare both groups (vitamin D and No vitamin D).

Time to reach undetectable levels of SARS COV2 Infection.

Time of normalization of symptoms and clinical parameters.

Time of normalization of radiological images.

Time of normalization of biochemical markers.

Time of normalization of molecular inflammatory markers.

Transfer to the Intensive care Unit.

Mortality rate.

ELIGIBILITY:
Inclusion Criteria:

* > 18 year
* Diagnosis of COVID-19
* Accept to participate in the study ( consent)

Exclusion Criteria:

* Pregnancy
* Allergy to vitamin D
* Consumption of any form of vitamin D during the last 3 months
* Expected fatal outcome in the next 24 hours
* Cognitive deterioration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-04-04 (Actual); Primary Completion 2020-09-14 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | Time to death or hospital discharge in days (average 12 days)
  Percentage of patients dying during hospitalization
Admission to Intensive Care Unit (ICU) | Time from hospital admission to discharge in days (average 12 days)
  Percentage of patients admitted to ICU and time in ICU
Time of hospitalization | Time of hospitalization in days (average 12 days)
  Number of days from hospital admission to discharge
Clinical changes | At the time of hospital admission and discharge (average 12 days)
  Percentage of patients with symptoms after treatment (Cough, fever, headache, weakness, dyspnoea, anosmia, diarrhoea, ageusia, others ...)
Radiological changes | At the time of hospital admission and discharge (average 12 days)
  Changes in the percentage of patients with radiological findings of pneumonia and severity
Calcidiol changes | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Calcidiol levels in ng/mL.
Inflammation markers changes (CRP) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  C-reactive protein (CRP) in mg/L
Inflammation markers changes (IL-6) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Interleukin-6 (IL-6) in pg/mL
Inflammation markers changes (Leucocytes) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Leucocytes in cells per liter
Inflammation markers changes (D-dimer) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  D-dimer in µg/mL
General biochemical parameters changes (Creatinine) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Creatinine in mg/dL
General biochemical parameters changes (Ferritin) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Ferritin in µg/L
General biochemical parameters changes (Bilirubin) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Bilirubin in mg/dL
General biochemical parameters changes (Albumin) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Albumin in g/dL
General biochemical parameters changes (Haemoglobin) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Haemoglobin in g/dL
General biochemical parameters changes (HDL cholesterol) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  High density lipoprotein (HDL cholesterol) in mg/dL
General biochemical parameters changes (Procalcitonin) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Procalcitonin in ng/mL
General biochemical parameters changes (Protonin) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Protonin in ng/L
General biochemical parameters changes (Calcium) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Calcium in mg/dL
General biochemical parameters changes (Phosphate) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  Phosphate in mg/dL
General biochemical parameters changes (pO2) | At the time of hospital admission (before initiation of treatment) and at hospital discharge (average 12 days)
  pO2 in mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cannata-Andia JB, Diaz-Sottolano A, Fernandez P, Palomo-Antequera C, Herrero-Puente P, Mouzo R, Carrillo-Lopez N, Panizo S, Ibanez GH, Cusumano CA, Ballarino C, Sanchez-Polo V, Pefaur-Penna J, Maderuelo-Riesco I, Calvino-Varela J, Gomez MD, Gomez-Alonso C, Cunningham J, Naves-Diaz M, Douthat W, Fernandez-Martin JL; COVID-VIT-D trial collaborators. A single-oral bolus of 100,000 IU of cholecalciferol at hospital admission did not improve outcomes in the COVID-19 disease: the COVID-VIT-D-a randomised multicentre international clinical trial. BMC Med. 2022 Feb 18;20(1):83. doi: 10.1186/s12916-022-02290-8. PMID 35177066